CLINICAL TRIAL: NCT02912572
Title: A Phase 2, Two-Group, Two-Stage, Open-Label Study of Avelumab in Patients With MSS, MSI-H and POLE-mutated Recurrent or Persistent Endometrial Cancer, Avelumab / Talazoparib in Patients With MSS Recurrent or Persistent Endometrial Cancer, and Avelumab / Axitinib in Patients With MSS Recurrent or Persistent Endometrial Cancer
Brief Title: Avelumab in Patients With MSS, MSI-H and POLE-mutated Recurrent or Persistent Endometrial Cancer and of Avelumab/Talazoparib and Avelumab/Axitinib in Patients With MSS Recurrent or Persistent Endometrial Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Panagiotis Konstantinopoulos, MD, PhD, MD, PhD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-322
Record Dates: First submitted 2016-09-20; First posted 2016-09-23 (Estimated); Results first posted 2024-07-05 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Endometrial Cancer
Keywords: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — avelumab; talazoparib; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pole Mutated Endometrial Cancer (Experimental): Participants with Pole mutated endometrial cancer Avelumab will be administered intravenously twice per cycle
  Interventions: Drug: Avelumab
- MSS Endometrial Cancer (Experimental): Participants with MSS mutated endometrial cancer Avelumab will be administered intravenously twice per cycle
  Interventions: Drug: Avelumab
- MSS Avelumab/Talazoparib Combination Arm (Experimental): Participants with MSS mutated endometrial cancer Avelumab will be administered intravenously twice per cycle Talazoparib will be administered one time per day by mouth
  Interventions: Drug: Avelumab; Drug: Talazoparib
- MSS Avelumab/Axitinib Combination Arm (Experimental): Participants with MSS mutated endometrial cancer Avelumab will be administered intravenously twice per cycle Axitinib will be administered twice per day by mouth
  Interventions: Drug: Avelumab; Drug: Axitinib

INTERVENTIONS:
Drug: Avelumab — Avelumab will be administered intravenously twice per cycle Each Cycle lasts 28 days Premedication Antihistamine and Paracetamol will be administered prior to treatment
Drug: Talazoparib — Talazoparib will be taken one time per day by mouth Each Cycle lasts 28 days
  Arms: MSS Avelumab/Talazoparib Combination Arm
Drug: Axitinib — Axitinib will be taken twice per day by mouth Each Cycle lasts 28 days
  Arms: MSS Avelumab/Axitinib Combination Arm

SUMMARY:
This research study is evaluating a drug called Avelumab alone and in combination with Talazoparib or Axitinib as a possible treatment for recurrent or metastatic endometrial cancer.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the effectiveness of an investigational drug to learn whether the drug works in treating a specific cancer. "Investigational" means that the drug is still being studied and that research doctors are trying to find out more about it-such as the safest dose to use, the side effects it may cause, and if the drug is effective for treating different types of cancer. It also means that the FDA (the U.S. Food and Drug Administration) has not yet approved the drug for use in patients, including people with Metastatic Endometrial Cancer.

Avelumab is a drug that may stop cancer cells from growing by enabling the activation of the immune system. Avelumab blocks an immune inhibiting signal that can impair the ability of the immune system to attack cancers.

Talazoparib is a drug that stops the activity of a protein (called PARP) that's involved in repairing damage to the DNA within your cells. When PARP is turned off by Talazoparib in cancer cells, DNA damage cannot be repaired and leads to the death of the cancer cells.

Axitinib is a drug that may stop cancer cells from growing by blocking certain proteins that cancer cells use to form new blood vessels, which the cancer needs in order to grow.

In this research study, the investigators are looking to see whether Avelumab, the combination of Avelumab and Talazoparib, or the combination of Avelumab and Axitinib are effective in treating recurrent and Metastatic Endometrial Cancer.

Additionally, the investigators are looking to see if participants whose tumors contain a particular genetic make-up will have better response to Avelumab, the combination of Avelumab and Talazoparib, or the combination of Avelumab and Axitinib.

ELIGIBILITY:
Inclusion Criteria:

Participants must be classified into one of the following cohorts of recurrent or persistent endometrial cancer of any histology:

The MSI/POLE cohort includes endometrial cancers that are:

--MSI-H as determined by immunohistochemical complete loss of expression (absence of nuclear immunoreactivity) of at least one of the mismatch repair genes MSH2, MSH6, MLH1 and PMS2. This test is now done routinely for every newly diagnosed endometrial cancer patient in most centers in the US.

And/OR:

--POLE-mutated, i.e. endometrial cancers known to harbor mutations in the exonuclease domain (amino acid residues 268-471) of polymerase e (POLE) as determined by targeted sequencing or other next generation sequencing assay. Any Clinical Laboratory Improvement Amendments (CLIA)-approved genomic test documenting mutations in the exonuclease domain of POLE gene (amino acid residues 268-471) in the tumor will be accepted as proof of presence of POLE mutations and will lead to classification into this patient cohort.

The MSS cohorts include:

* Endometrial cancers that are MSS as determined by normal immunohistochemical nuclear expression of all the mismatch repair genes MSH2, MSH6, MLH1 and PMS2. Tumors which have not been sequenced for POLE mutations (i.e. their POLE mutations status is unknown) but are MSS, will be included in this cohort.

  * All patients must have measurable disease as defined by RECIST 1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be >= 10 mm when measured by CT, MRI or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray. Lymph nodes must be > 15 mm in short axis when measured by CT or MRI.
  * Prior Therapy:
* There is no upper limit of prior therapies but patients must have had one prior chemotherapeutic regimen for management of endometrial carcinoma. Initial treatment may include chemotherapy, chemotherapy and radiation therapy, and/or consolidation/maintenance therapy. Any platinum based chemotherapy (single agent platinum or any platinum doublet) administered in conjunction with primary radiation as a radio-sensitizer WILL be counted as a systemic chemotherapy regimen. Furthermore, patients who have only received chemotherapy in the adjuvant setting will be eligible for the study.
* Prior hormonal therapy is allowed.
* Patients must NOT have received any class of drugs targeted to the PD-1/PD-L1 pathway.
* Patients must NOT have received any prior PARP inhibitor therapy (for patients being considered for the avelumab/talazoparib cohort only).
* Patients must NOT have received prior axitinib (for patients being considered for the avelumab/axitinib cohort only).

  * Age of 18 or greater years. Because insufficient dosing or adverse event data are currently available on the use of Avelumab, talazoparib, and/or axitinib in participants < 18 years of age, children are excluded from the study. Endometrial cancer is very rare in the pediatric population.
  * ECOG performance status 0 or 1 (reference Appendix A for ECOG performance status criteria).
  * Availability of a formalin fixed paraffin embedded (FFPE) block of cancer tissue OR 15 unstained 5-micron slides from the original surgery or biopsy or from a biopsy of recurrent disease.
  * Participants must have normal organ and marrow function as defined below:
* absolute neutrophil count >1,500/mcL
* platelets >100,000/mcL
* hemoglobin ≥ 9g/dL
* total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
* creatinine within normal institutional limits OR
* creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.

Please note: creatinine clearance (CLCR) should be estimated according to the Cockcroft-Gault formula as:

CLCR={[(140-age) × weight)]/(72 x SCR)} × 0.85 where CLCR (creatinine clearance) is measured in mL/min, age is expressed in years, weight in kilograms (kg), and SCR (serum creatinine) in mg/dL.

NOTE: Patients with moderate renal impairment (defined as an estimated creatinine clearance of 30-59 mL/min) will receive a reduced starting dose of Talazoparib at 0.75 mg PO QD.

* Participant must not be pregnant or breastfeeding given that avelumab is an agent with unknown effects in pregnancy and breastfeeding and the potential for teratogenesis. Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or post-menopausal (defined as ≥ 12 months with no menses without an alternative medical cause). Serum pregnancy test (for females of childbearing potential) negative at screening.
* The effects of avelumab on the developing human fetus are unknown. For this reason and because some immunomodulatory agents are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Toxicities of prior therapy (excepting alopecia and sensory neuropathy) should be resolved to < grade 2 per the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4. All appropriate treatment areas should have access to a copy of the CTCAE version 4. A copy of the CTCAE version 4 can be downloaded from the CTEP website at: http://ctep.cancer.gov.
* Ability to understand and the willingness to sign a written informed consent document.

Additional inclusion criteria for the avelumab/axitinib cohort:

* Participants must have adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as systolic BP that must be ≤140 mmHg and diastolic BP that must be ≤90 mmHg on two separate BP readings taken at least 1 hour apart at screening.
* Participants must have LVEF ≥ lower limit of normal (LLN) as assessed by either multigated acquisition (MUGA) scan or echocardiogram (ECHO).

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants who are receiving any other investigational agents.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to avelumab or any component in its formulations, or compounds of similar chemical or biologic composition to avelumab. Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3 NCI CTCAE v 4.03), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma)
* Participants with a history of treatment with an anti-PD-1, anti-PD-L1, anti-CTLA-4 or other investigational agents that target immune checkpoint inhibitors.
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness, which may compromise the efficacy of immunostimulatory therapy.
* Positive test for HBV surface antigen
* Positive Hepatitis C antibody and positive confirmatory HCV RNA test. The confirmatory HCV RNA test is not required if the HCV antibody is negative. If Hepatitis C antibody is positive, the confirmatory HCV RNA test should be done and if it is negative, then participants are eligible.
* Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg or 10 mg equivalent prednisone per day
* Active infection requiring systemic therapy.
* Current or prior use of immunosuppressive medication within 7 days prior to enrollment with the following exceptions to this exclusion criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection);
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent;
  * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
* Prior organ transplantation including allogeneic stem-cell transplantation.
* Severe gastrointestinal conditions such as clinical or radiological evidence of bowel obstruction within 4 weeks prior to study entry, uncontrolled diarrhea in the last 4 weeks prior to enrollment, or history of inflammatory bowel disease.
* Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Known alcohol or drug abuse.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: breast cancer in situ, cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* All other significant diseases (for example, inflammatory bowel disease, uncontrolled asthma), which, in the opinion of the Investigator, might impair the subject's tolerance of trial treatment.
* Any psychiatric condition that would prohibit the understanding or rendering of informed consent
* Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines.
* Patients may not use natural herbal products or other "folk remedies" while participating in this study. Herbal medications include, but are not limited to St. John's Wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng.

Additional exclusion criteria for the avelumab/axitinib cohort:

* Participants having >1+ proteinuria on urinalysis or UPCR >1 will undergo a 24-hour urine collection for quantitative assessment of proteinuria. Participants with urine protein >1 g/24-hours will be ineligible.
* Participants with concern for bowel or serosal involvement will be ineligible, due to the risk of perforation or fistulization with anti-angiogenic agents.
* Participants will be ineligible if they have active gastrointestinal bleeding, as evidenced by clinically significant hematemesis, hematochezia, or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy.
* Participants will be ineligible if using anticoagulant therapy with oral vitamin K antagonists, novel oral anticoagulants (NOACs), or direct oral anticoagulants (DOACs), inclusive of direct thrombin inhibitors and direct factor Xa inhibitors. Therapeutic use of low molecular weight heparin is allowed. Low dose heparin required for maintenance of patency of central venous access devices are allowed.
* Grade ≥3 hemorrhage within 4 weeks preceding Cycle 1 Day 1 treatment.
* Ongoing cardiac dysrhythmias of CTCAE Grade≥2, or prolongation of the QTc interval to >500 msec
* Current use or anticipated need for treatment with drugs or foods that are known to be either:

  * Strong CYP3A4/5 inhibitors, including administration within 10 days prior to Cycle 1 Day 1 treatment, including but not limited to grapefruit juice, grapefruit-related fruits (Seville oranges, pomelos), ketoconazole, miconazole, itraconazole, voriconazole, posaconazole, clarithromycin, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, amprenavir, fosamprenavir nefazodone, lopinavir, troleandomycin, mibefradil, conivaptan. The topical use of these medications is allowed if systemic absorption is considered minimal.
  * Strong CYP3A4/5 inducers, including administration within 10 days prior to Cycle 1 Day 1 treatment, including but not limited to phenobarbital, rifampin, phenytoin, carbamazepine, rifabutin, rifapentine, clevidipine, St. John's wort.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2026-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Konstantinopoulos, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Konstantinopoulos PA, Gockley AA, Xiong N, Krasner C, Horowitz N, Campos S, Wright AA, Liu JF, Shea M, Yeku O, Castro C, Polak M, Lee EK, Sawyer H, Bowes B, Moroney J, Cheng SC, Tayob N, Bouberhan S, Spriggs D, Penson RT, Fleming GF, Nucci MR, Matulonis UA. Evaluation of Treatment With Talazoparib and Avelumab in Patients With Recurrent Mismatch Repair Proficient Endometrial Cancer. JAMA Oncol. 2022 Sep 1;8(9):1317-1322. doi: 10.1001/jamaoncol.2022.2181. PMID 35900726

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 106 participants who enrolled in the study, 5 participants never started treatment and were excluded from the study: two participants were excluded from the intervention due to not re-meeting eligibility parameters prior to treatment initiation, two participants were hospitalized prior to group assignment and never re-screened for the study, and one participant was excluded from the study per provider discretion. Therefore, 101 participants started on study.
Groups:
- MSI-H/POLE-Mutated Avelumab Arm: Participants with MSI-H and/or POLE-mutated endometrial cancer received Avelumab at 10 mg/kg intravenously on Day 1 and Day 15 of each 28-day cycle.
- MSS Avelumab Arm: Participants with MSS endometrial cancer received Avelumab at 10 mg/kg intravenously on Day 1 and Day 15 of each 28-day cycle.
- MSS Avelumab/Talazoparib Combination Arm: Participants with MSS endometrial cancer received Avelumab at 10 mg/kg intravenously on Day 1 and Day 15 of each 28-day cycle in combination with 1mg Talazoparib orally once daily.
- MSS Avelumab/Axitinib Combination Arm: Participants with MSS endometrial cancer received Avelumab at 800mg intravenously on Day 1 and Day 15 of each 28-day cycle in combination with 5mg Axitinib orally twice daily.
Period: Overall Study
Arm/Group | MSI-H/POLE-Mutated Avelumab Arm | MSS Avelumab Arm | MSS Avelumab/Talazoparib Combination Arm | MSS Avelumab/Axitinib Combination Arm
Started | 15 | 16 | 35 | 35
Completed | 15 | 16 | 35 | 35
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MSI-H/POLE-Mutated Avelumab Arm | MSS Avelumab Arm | MSS Avelumab/Talazoparib Combination Arm | MSS Avelumab/Axitinib Combination Arm | Total
Number analyzed (Participants) | 15 | 16 | 35 | 35 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (6.98) | 65.9 (8.41) | 67.9 (8.41) | 65.1 (9.23) | 65.9 (8.81)
Age, Customized [Median (Full Range); unit: years] | 63.7 [52.4 to 76.4] | 66.5 [42.0 to 82.4] | 68.8 [43.7 to 88.1] | 65.5 [28.1 to 80.2] | 66.1 [28.1 to 88.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 35 | 35 | 101
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 14 | 13 | 23 | 31 | 81
  Unknown or Not Reported | 1 | 3 | 12 | 2 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 5 | 10 | 17
  White | 13 | 13 | 18 | 22 | 66
  More than one race | 0 | 0 | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 11 | 2 | 15
Stage at Diagnosis [Count of Participants; unit: Participants] — Staging was based on the FIGO (International Federation of Gynecology and Obstetrics) system. Stage I cancers usually have not grown deeply into nearby tissues. Stage II and III cancers have grown more deeply into nearby tissue and may have spread to lymph nodes. Stage IV cancers have spread to other organs or parts of the body. Higher stages are typically associated with worse outcomes.
  Participants
    Stage I | 8 | 5 | 9 | 6 | 28
    Stage II | 2 | 1 | 3 | 1 | 7
    Stage III | 4 | 3 | 6 | 12 | 25
    Stage IV | 1 | 7 | 17 | 16 | 41
Histology [Count of Participants; unit: Participants]
  Endometrioid | 14 | 6 | 11 | 11 | 42
  Mixed | 1 | 3 | 5 | 0 | 9
  Clear Cell | 0 | 0 | 3 | 4 | 7
  Carcinosarcoma | 0 | 2 | 4 | 5 | 11
  Serous | 0 | 3 | 12 | 15 | 30
  Adenocarcinoma not otherwise specified | 0 | 2 | 0 | 0 | 2
Number of Prior Lines of Therapy [Count of Participants; unit: Participants]
  1 | 6 | 3 | 10 | 27 | 46
  2 | 3 | 6 | 3 | 3 | 15
  3+ | 6 | 7 | 22 | 5 | 40

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The objective response rate was determined by the frequency of patients who had objective tumor response, determined per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI, where objective response represents either a confirmed complete response (CR; disappearance of all target lesions) or a confirmed partial response (PR; at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum diameters); objective response = CR + PR.
Time Frame: Up to 39 months
Measure: Count of Participants; unit: Participants
Arm/Group | MSI-H/POLE-Mutated Avelumab Arm | MSS Avelumab Arm | MSS Avelumab/Talazoparib Combination Arm | MSS Avelumab/Axitinib Combination Arm
Number analyzed (Participants) | 15 | 16 | 35 | 35
Participants | 4 | 1 | 4 | 9

2. Primary Outcome: Progression-Free Survival at 6 Months
Description: Progression-free survival at 6 months was determined by the frequency of patients who survived progression-free for at least 6 months after initiating study treatment by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), where disease progression represents at least a 20% increase in the sum of diameters of target lesions, appearance of one or more new lesions, or unequivocal progression of existing non-target lesions.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | MSI-H/POLE-Mutated Avelumab Arm | MSS Avelumab Arm | MSS Avelumab/Talazoparib Combination Arm | MSS Avelumab/Axitinib Combination Arm
Number analyzed (Participants) | 15 | 16 | 35 | 35
Participants | 6 | 1 | 8 | 14

3. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival was determined per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), where disease progression represents at least a 20% increase in the sum of diameters of target lesions, appearance of one or more new lesions, or unequivocal progression of existing non-target lesions. The distribution of progression-free times will be estimated using Kaplan-Meier analysis.
Time Frame: Interval from start of treatment to documented disease progression per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death from any cause, whichever occurs first.
Reporting Status: Not Posted, anticipated posting 2027-11

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from registration to death due to any cause, or censored at date last known alive. The distribution of overall survival times will be estimated using Kaplan-Meier analysis.
Time Frame: Participants are followed for survival status from registration through up to 3 years after removal from study intervention
Reporting Status: Not Posted, anticipated posting 2027-11

5. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Description: As classified by the common terminology criteria for adverse events (CTCAE) version 4.0
Time Frame: Adverse event data was collected for all participants through 30 days after last intervention
Reporting Status: Not Posted, anticipated posting 2027-11

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for all participants through 30 days after last intervention (up to 85 months).
Arm/Group | MSI-H/POLE-Mutated Avelumab Arm | MSS Avelumab Arm | MSS Avelumab/Talazoparib Combination Arm | MSS Avelumab/Axitinib Combination Arm
All-Cause Mortality (participants affected / at risk) | 0/15 | 3/16 | 0/35 | 1/35
Serious Adverse Events (participants affected / at risk) | 4/15 | 7/16 | 11/35 | 16/35
Other Adverse Events (participants affected / at risk) | 15/15 | 15/16 | 35/35 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MSI-H/POLE-Mutated Avelumab Arm (N=15) | MSS Avelumab Arm (N=16) | MSS Avelumab/Talazoparib Combination Arm (N=35) | MSS Avelumab/Axitinib Combination Arm (N=35)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Aortic valve disease (Cardiac disorders) | 0 | 1 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 0 | 2
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1
Eye disorders - Other, specify (Hemianopsia) (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Jejunal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 2 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Death NOS (General disorders) | 0 | 2 | 0 | 0
General disorders and administration site conditions - Other, specify (Failure to thrive) (General disorders) | 0 | 0 | 1 | 0
Infusion related reaction (General disorders) | 0 | 0 | 1 | 1
Infections and infestations - Other (Infections and infestations) | 1 | 0 | 0 | 0
Infections and infestations - Other, specify (Influenza A) (Infections and infestations) | 0 | 1 | 0 | 0
Infections and infestations - Other, specify (Influenza B) (Infections and infestations) | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Metabolism and nutrition disorders - Other, specify (Failure to thrive) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 3
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal and urinary disorders - Other, specify (Bilateral hydronephrosis) (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hematoma (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 4
Thromboembolic event (Vascular disorders) | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MSI-H/POLE-Mutated Avelumab Arm (N=15) | MSS Avelumab Arm (N=16) | MSS Avelumab/Talazoparib Combination Arm (N=35) | MSS Avelumab/Axitinib Combination Arm (N=35)
Grade 1-2 Anemia (Blood and lymphatic system disorders) | 6 | 5 | 9 | 8
Grade 1-2 Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Grade 1-2 Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Grade 3 Anemia (Blood and lymphatic system disorders) | 4 | 0 | 16 | 1
Grade 3 Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Grade 4 Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Grade 1-2 Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 0 | 2
Grade 1-2 Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Grade 1-2 Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 1
Grade 1-2 Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1
Grade 1-2 Sinus bradycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Grade 1-2 Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 3
Grade 1-2 Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Grade 3 Aortic valve disease (Cardiac disorders) | 0 | 1 | 0 | 0
Grade 3 Heart failure (Cardiac disorders) | 0 | 0 | 0 | 1
Grade 3 Restrictive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Grade 3 Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Grade 1-2 Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Grade 1-2 Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Grade 1-2 Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Grade 1-2 Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Grade 1-2 Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Grade 1-2 Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0
Grade 1-2 Endocrine disorders - Other (Endocrine disorders) | 0 | 1 | 0 | 1
Grade 1-2 Hyperthyroidism (Endocrine disorders) | 2 | 1 | 1 | 4
Grade 1-2 Hypothyroidism (Endocrine disorders) | 3 | 1 | 4 | 11
Grade 3 Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Grade 1-2 Blurred vision (Eye disorders) | 0 | 0 | 1 | 2
Grade 1-2 Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0
Grade 1-2 Dry eye (Eye disorders) | 1 | 0 | 2 | 1
Grade 1-2 Eye disorders - Other (Eye disorders) | 1 | 0 | 1 | 1
Grade 1-2 Eye pain (Eye disorders) | 0 | 0 | 2 | 0
Grade 1-2 Uveitis (Eye disorders) | 0 | 0 | 1 | 0
Grade 1-2 Vitreous hemorrhage (Eye disorders) | 0 | 1 | 1 | 0
Grade 1-2 Watering eyes (Eye disorders) | 0 | 0 | 0 | 1
Grade 3 Eye disorders - Other (Eye disorders) | 0 | 1 | 0 | 0
Grade 1-2 Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Grade 1-2 Abdominal pain (Gastrointestinal disorders) | 5 | 4 | 7 | 17
Grade 1-2 Ascites (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Grade 1-2 Bloating (Gastrointestinal disorders) | 0 | 1 | 2 | 5
Grade 1-2 Colitis (Gastrointestinal disorders) | 2 | 1 | 1 | 1
Grade 1-2 Constipation (Gastrointestinal disorders) | 5 | 1 | 7 | 13
Grade 1-2 Diarrhea (Gastrointestinal disorders) | 7 | 2 | 9 | 20
Grade 1-2 Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 4
Grade 1-2 Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Grade 1-2 Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Grade 1-2 Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Grade 1-2 Esophageal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Grade 1-2 Fecal incontinence (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Grade 1-2 Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Grade 1-2 Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 3
Grade 1-2 Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0 | 3 | 1
Grade 1-2 Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Grade 1-2 Hemorrhoids (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Grade 1-2 Jejunal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Grade 1-2 Jejunal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Grade 1-2 Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Grade 1-2 Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 2 | 8
Grade 1-2 Nausea (Gastrointestinal disorders) | 6 | 4 | 16 | 18
Grade 1-2 Oral dysesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Grade 1-2 Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Grade 1-2 Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 5
Grade 1-2 Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Grade 1-2 Rectal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Grade 1-2 Tooth development disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Grade 1-2 Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Grade 1-2 Vomiting (Gastrointestinal disorders) | 5 | 4 | 7 | 13
Grade 3 Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Grade 3 Anal mucositis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Grade 3 Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Grade 3 Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Grade 3 Diarrhea (Gastrointestinal disorders) | 3 | 0 | 0 | 2
Grade 3 Gastric hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Grade 3 Jejunal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Grade 3 Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Grade 3 Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 2 | 1
Grade 3 Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Grade 3 Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Grade 4 Gastric perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Grade 1-2 Chills (General disorders) | 3 | 3 | 3 | 6
Grade 1-2 Edema face (General disorders) | 0 | 0 | 1 | 0
Grade 1-2 Edema limbs (General disorders) | 2 | 1 | 7 | 10
Grade 1-2 Edema trunk (General disorders) | 0 | 0 | 0 | 1
Grade 1-2 Facial pain (General disorders) | 0 | 1 | 0 | 0
Grade 1-2 Fatigue (General disorders) | 7 | 7 | 15 | 21
Grade 1-2 Fever (General disorders) | 3 | 2 | 3 | 3
Grade 1-2 Flu like symptoms (General disorders) | 1 | 1 | 0 | 4
Grade 1-2 Gait disturbance (General disorders) | 0 | 1 | 1 | 1
Grade 1-2 General disorders and administration site conditions - Other (General disorders) | 1 | 1 | 1 | 7
Grade 1-2 Infusion related reaction (General disorders) | 0 | 3 | 3 | 2
Grade 1-2 Irritability (General disorders) | 0 | 0 | 0 | 1
Grade 1-2 Malaise (General disorders) | 0 | 0 | 2 | 0
Grade 1-2 Non-cardiac chest pain (General disorders) | 2 | 1 | 0 | 6
Grade 1-2 Pain (General disorders) | 5 | 3 | 1 | 8
Grade 3 Edema face (General disorders) | 0 | 0 | 0 | 1
Grade 3 Fatigue (General disorders) | 1 | 0 | 4 | 2
Grade 3 Flu like symptoms (General disorders) | 1 | 0 | 0 | 0
Grade 3 General disorders and administration site conditions - Other (General disorders) | 0 | 0 | 1 | 0
Grade 3 Infusion related reaction (General disorders) | 0 | 0 | 1 | 2
Grade 3 Pain (General disorders) | 1 | 0 | 0 | 0
Grade 1-2 Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Grade 1-2 Conjunctivitis infective (Infections and infestations) | 1 | 0 | 0 | 0
Grade 1-2 Eye infection (Infections and infestations) | 1 | 0 | 0 | 0
Grade 1-2 Infections and infestations - Other (Infections and infestations) | 3 | 1 | 2 | 5
Grade 1-2 Lung infection (Infections and infestations) | 0 | 1 | 2 | 0
Grade 1-2 Mucosal infection (Infections and infestations) | 0 | 0 | 1 | 1
Grade 1-2 Papulopustular rash (Infections and infestations) | 0 | 0 | 0 | 1
Grade 1-2 Paronychia (Infections and infestations) | 0 | 0 | 0 | 1
Grade 1-2 Rash pustular (Infections and infestations) | 0 | 0 | 0 | 1
Grade 1-2 Sinusitis (Infections and infestations) | 0 | 1 | 3 | 0
Grade 1-2 Skin infection (Infections and infestations) | 3 | 0 | 0 | 1
Grade 1-2 Tooth infection (Infections and infestations) | 1 | 1 | 0 | 0
Grade 1-2 Upper respiratory infection (Infections and infestations) | 4 | 2 | 2 | 2
Grade 1-2 Urinary tract infection (Infections and infestations) | 2 | 2 | 2 | 8
Grade 1-2 Vulval infection (Infections and infestations) | 0 | 1 | 0 | 0
Grade 1-2 Wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Grade 3 Infections and infestations - Other (Infections and infestations) | 1 | 1 | 0 | 0
Grade 3 Kidney infection (Infections and infestations) | 1 | 0 | 0 | 0
Grade 3 Lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Grade 3 Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Grade 1-2 Bruising (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 4
Grade 1-2 Fall (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 3
Grade 1-2 Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Grade 1-2 Injury to jugular vein (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Grade 1-2 Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Grade 1-2 Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Grade 1-2 Alanine aminotransferase increased (Investigations) | 3 | 0 | 4 | 11
Grade 1-2 Alkaline phosphatase increased (Investigations) | 1 | 1 | 1 | 2
Grade 1-2 Aspartate aminotransferase increased (Investigations) | 4 | 1 | 5 | 10
Grade 1-2 Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 2
Grade 1-2 Cardiac troponin I increased (Investigations) | 0 | 0 | 0 | 2
Grade 1-2 Cholesterol high (Investigations) | 0 | 0 | 0 | 1
Grade 1-2 Creatinine increased (Investigations) | 1 | 2 | 5 | 1
Grade 1-2 Hemoglobin increased (Investigations) | 0 | 0 | 0 | 2
Grade 1-2 INR increased (Investigations) | 0 | 0 | 1 | 0
Grade 1-2 Investigations - Other (Investigations) | 1 | 1 | 2 | 2
Grade 1-2 Lymphocyte count decreased (Investigations) | 2 | 1 | 0 | 4
Grade 1-2 Neutrophil count decreased (Investigations) | 3 | 2 | 8 | 3
Grade 1-2 Platelet count decreased (Investigations) | 4 | 1 | 15 | 3
Grade 1-2 Serum amylase increased (Investigations) | 0 | 0 | 0 | 1
Grade 1-2 Urine output decreased (Investigations) | 1 | 0 | 0 | 0
Grade 1-2 Weight loss (Investigations) | 0 | 0 | 1 | 4
Grade 1-2 White blood cell decreased (Investigations) | 3 | 0 | 4 | 0
Grade 3 Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2
Grade 3 Alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 1
Grade 3 Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2
Grade 3 Creatinine increased (Investigations) | 0 | 0 | 1 | 0
Grade 3 Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0
Grade 3 Neutrophil count decreased (Investigations) | 0 | 0 | 4 | 0
Grade 3 Platelet count decreased (Investigations) | 0 | 0 | 7 | 0
Grade 4 Platelet count decreased (Investigations) | 0 | 0 | 3 | 0
Grade 1-2 Anorexia (Metabolism and nutrition disorders) | 2 | 3 | 7 | 18
Grade 1-2 Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Grade 1-2 Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1
Grade 1-2 Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2 | 2 | 3
Grade 1-2 Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Grade 1-2 Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Grade 1-2 Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Grade 1-2 Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Grade 1-2 Hypokalemia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 6
Grade 1-2 Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 13
Grade 1-2 Hyponatremia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 4
Grade 1-2 Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Grade 1-2 Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Grade 3 Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Grade 3 Hypokalemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0
Grade 3 Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 2
Grade 3 Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Grade 3 Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Grade 3 Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Grade 1-2 Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4 | 5
Grade 1-2 Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Grade 1-2 Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 5 | 8
Grade 1-2 Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Grade 1-2 Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Grade 1-2 Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Grade 1-2 Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Grade 1-2 Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 4
Grade 1-2 Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Grade 1-2 Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Grade 1-2 Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 3
Grade 1-2 Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5 | 6
Grade 1-2 Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Grade 1-2 Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Grade 1-2 Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | 3
Grade 3 Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Grade 3 Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Grade 3 Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Grade 3 Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Grade 3 Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Grade 3 Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Grade 3 Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Grade 3 Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Grade 1-2 Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Grade 1-2 Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Grade 1-2 Dizziness (Nervous system disorders) | 2 | 1 | 5 | 13
Grade 1-2 Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 6
Grade 1-2 Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Grade 1-2 Headache (Nervous system disorders) | 5 | 1 | 5 | 12
Grade 1-2 Nervous system disorders - Other (Nervous system disorders) | 0 | 0 | 2 | 2
Grade 1-2 Paresthesia (Nervous system disorders) | 1 | 1 | 1 | 2
Grade 1-2 Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Grade 1-2 Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 4 | 3
Grade 1-2 Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Grade 1-2 Sinus pain (Nervous system disorders) | 0 | 1 | 0 | 1
Grade 1-2 Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Grade 1-2 Tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Grade 3 Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Grade 3 Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Grade 3 Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Grade 3 Vasovagal reaction (Nervous system disorders) | 0 | 1 | 0 | 0
Grade 1-2 Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 3
Grade 1-2 Depression (Psychiatric disorders) | 3 | 0 | 2 | 3
Grade 1-2 Insomnia (Psychiatric disorders) | 1 | 0 | 2 | 1
Grade 3 Confusion (Psychiatric disorders) | 0 | 0 | 0 | 1
Grade 1-2 Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 1
Grade 1-2 Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 0 | 0
Grade 1-2 Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 5
Grade 1-2 Proteinuria (Renal and urinary disorders) | 0 | 0 | 2 | 9
Grade 1-2 Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 0 | 0 | 3
Grade 1-2 Urinary frequency (Renal and urinary disorders) | 1 | 0 | 0 | 3
Grade 1-2 Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Grade 1-2 Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 2
Grade 1-2 Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Grade 1-2 Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 1 | 3
Grade 3 Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 2
Grade 3 Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0
Grade 3 Hematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Grade 3 Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Grade 3 Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 1 | 0 | 0
Grade 3 Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 3 | 1
Grade 1-2 Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 2 | 4
Grade 1-2 Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Grade 1-2 Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1 | 2 | 0 | 1
Grade 1-2 Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 2
Grade 1-2 Vaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Grade 1-2 Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 2 | 3
Grade 1-2 Vaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Grade 1-2 Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Grade 1-2 Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Grade 1-2 Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 5 | 7
Grade 1-2 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 5 | 13
Grade 1-2 Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3
Grade 1-2 Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Grade 1-2 Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 6
Grade 1-2 Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Grade 1-2 Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 6
Grade 1-2 Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Grade 1-2 Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Grade 1-2 Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Grade 1-2 Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Grade 1-2 Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Grade 1-2 Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Grade 1-2 Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Grade 1-2 Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 1
Grade 1-2 Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Grade 1-2 Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Grade 1-2 Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 5
Grade 1-2 Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Grade 1-2 Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Grade 3 Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Grade 3 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Grade 3 Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Grade 4 Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Grade 1-2 Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 3
Grade 1-2 Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 6
Grade 1-2 Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Grade 1-2 Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Grade 1-2 Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Grade 1-2 Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 5
Grade 1-2 Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 5 | 2
Grade 1-2 Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Grade 1-2 Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 3 | 3
Grade 1-2 Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Grade 1-2 Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Grade 1-2 Skin/subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 6 | 1 | 3 | 8
Grade 1-2 Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Grade 3 Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Grade 3 Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Grade 1-2 Surgical and medical procedures - Other (Surgical and medical procedures) | 1 | 1 | 0 | 0
Grade 1-2 Flushing (Vascular disorders) | 1 | 0 | 0 | 1
Grade 1-2 Hematoma (Vascular disorders) | 1 | 2 | 0 | 1
Grade 1-2 Hypertension (Vascular disorders) | 2 | 2 | 2 | 10
Grade 1-2 Hypotension (Vascular disorders) | 0 | 1 | 0 | 3
Grade 1-2 Thromboembolic event (Vascular disorders) | 1 | 1 | 0 | 0
Grade 1-2 Vascular disorders - Other (Vascular disorders) | 1 | 0 | 0 | 0
Grade 3 Hypertension (Vascular disorders) | 1 | 1 | 1 | 13
Grade 3 Thromboembolic event (Vascular disorders) | 0 | 2 | 2 | 1
Grade 4 Hematoma (Vascular disorders) | 1 | 0 | 0 | 0
Grade 4 Hypertension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/72/NCT02912572/Prot_SAP_000.pdf